CLINICAL TRIAL: NCT00115830
Title: Rho Kinase in Patients With Atherosclerosis: Effects of Statins - A Double Blind, Randomized Clinical Trial Comparing Rosuvastatin and Atorvastatin
Brief Title: Rho Kinase in Patients With Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004P-002254
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atorvastatin
Drug: Rosuvastatin

SUMMARY:
The purpose of the study is to investigate the effects of atorvastatin (Lipitor) and rosuvastatin (Crestor), United States Food and Drug Administration (FDA) approved drugs commonly prescribed by doctors to lower cholesterol, on certain functions of platelets (cells that cause blood clots), white blood cells (cells that are responsible for inflammation), and blood flow regulation by arteries. This is important because we are looking at ways to more effectively prevent atherosclerosis (plaque buildup in blood vessels) and heart disease. Many studies have demonstrated that these drugs are effective at reducing inflammation and stabilizing plaques. We are interested in better understanding the effects of these medicines on inflammation (pain and swelling) and the mechanism by which they act.

Hypothesis: Atorvastatin (40mg) will reduce inflammatory markers and activity more than Rosuvastatin (10mg) in spite of equal LDL-C reduction.

DETAILED DESCRIPTION:
A double-blind controlled trial with two arms will be conducted at Brigham and Women's Hospital (BWH). We will screen subjects with stable atherosclerosis to complete enrollment of 40 subjects in the study (see inclusion and exclusion criteria section below). A central pharmacist at BWH will randomize the patients to 40mg of atorvastatin (n=20) or 10mg of rosuvastatin (n=20) for 28 days. If the patient is already on a statin a two-week washout period will be required prior to trial initiation. Our subjects, clinicians, data collectors, outcomes assessors and statisticians will be blind with regards to the patient allocation. There are a total of 3 visits for each patient: a short screening visit, an initial visit for baseline data (90 min.) and a final visit after 28 days. Our participants will be asked to take the medication every day at the same time between 9pm and 10pm. Each visit will take place between 7am and 9am. Patients will be instructed to fast overnight for a minimum of 8hrs. They will also be advised not to make any other changes to their current medications and lifestyle for 28 days while in the study and to record in a diary any side effects, missed doses, or changes in concomitant medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 40 to 80 years
* Documented stable atherosclerosis by angiography or vascular ultrasound (more that 20% luminal narrowing), previous myocardial infarction, ischemic stroke, peripheral arterial disease or type 2 diabetes mellitus (coronary heart disease (CHD) risk equivalent - Adult Treatment Program (ATP)-III guidelines)
* LDL-cholesterol >100mg/dL (indication to treat with statin)
* Written informed consent
* Primary care physician authorization letter to participate in the study.

Exclusion Criteria:

* Inability to give consent
* Pre-menopausal women
* Current use of antibiotics, anti-inflammatory or immunosuppressant drugs
* History of LFT >2 times the upper normal limit
* History of myopathy/myositis or CPK > 10 times the upper normal limit
* CPK above normal limits at study onset
* Any evidence of inflammatory, infectious or neoplastic disease
* History of CABG, PCI or acute ischemic syndrome in the preceding 3 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-12; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Selwyn, MD, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Womens Hospital, Boston, Massachusetts, United States